CLINICAL TRIAL: NCT02949362
Title: A Retrospective and Prospective, Open-label, Long-term Safety and Efficacy Study of Teduglutide in Pediatric Subjects With Short Bowel Syndrome Who Completed TED-C13-003
Brief Title: Long-term Study of Teduglutide in Pediatric Subjects With Short Bowel Syndrome Who Completed the TED-C13-003 Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHP633-303; 2016-000863-17 (EudraCT Number)
Record Dates: First submitted 2016-10-05; First posted 2016-10-31 (Estimated); Results first posted 2021-06-14 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome | interventions — teduglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Standard of Care (SOC) Treatment +/- Teduglutide (Experimental): TED 0.05mg/kg subcutaneous injections once daily as needed in addition to SOC treatment
  Interventions: Drug: Teduglutide; Other: SOC

INTERVENTIONS:
Drug: Teduglutide — 0.05mg/kg
Other: SOC — Standard safety assessments and adjustments in nutritional support will be provided for all subjects throughout the study, including any teduglutide treatment periods

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of teduglutide treatment of children with short bowel syndrome (SBS) who completed the TED-C13-003 study over a long-term period. It will evaluate how these children fared after the TED-C13-003 study ended. This study will also offer teduglutide treatment to eligible subjects, regardless of treatment received in TED-C13-003.

ELIGIBILITY:
Inclusion Criteria:

1. Subject provides written informed consent (subject, parent or legal guardian and, as appropriate, subject informed assent) to participate in the study before completing any study-related procedures.
2. Subject completed the TED-C13-003 study (including subjects in the standard of care treatment arm).
3. Subject understands and is willing and able to fully adhere to study requirements as defined in this protocol.

Exclusion Criteria:

There are no exclusion criteria for this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-12-09 (Actual); Primary Completion 2020-07-14 (Actual); Study Completion 2020-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shire Study Physician, Principal Investigator — Shire
Locations (11):
- United States (10):
  - Childrens Hospital Los Angeles - RHU, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Riley Hospital for Children, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Children's Hospital at Montefiore, The Bronx, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin
- Great Ormond Children's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as the data are subject to contractual (or consent) provisions that prohibit transfer to third parties.

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fd94db2bf003ab470b2

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed TED-C13-003 (NCT01952080) were enrolled in this study which was conducted at 11 sites in the United States and United Kingdom between 09 December 2016 (first participant first visit) and 14 July 2020 (last participant last visit).
Pre-assignment Details: A total of 29 participants were enrolled in this study, 29 participants consented to retrospective period. Of these, 24 enrolled into Retro TED/NTT (did not receive teduglutide) and 5 into Retro TED/TED (received teduglutide). Out of 29 participants of retrospective period, 24 enrolled into prospective period (ANY TED group), of these, 19 in TED/TED and 5 in TED/NTT.
Groups:
- Retrospective TED/NTT Group: Participants received teduglutide 0.05 milligrams per kilogram (mg/kg) subcutaneous injection once daily in TED-C13-003 (NCT01952080) and did not receive teduglutide in retrospective period in the current study SHP633-303.
- Retrospective TED/TED Group: Participants who received teduglutide 0.05 mg/kg subcutaneous injection once daily in TED-C13-003 (NCT01952080) and also received teduglutide in retrospective period in the current study SHP633-303.
- Prospective TED/NTT Group: Participants who received teduglutide 0.05 mg/kg subcutaneous injection once daily in TED-C13-003 (NCT01952080) and did not receive teduglutide in prospective period in the current study SHP633-303 up to 24 weeks.
- Prospective TED/TED Group: Participants who received teduglutide 0.05 mg/kg subcutaneous injection once daily in TED-C13-003 (NCT01952080) and also received teduglutide in prospective period in the current study SHP633-303 up to 24 weeks.
Period: Retrospective Period
Arm/Group | Retrospective TED/NTT Group | Retrospective TED/TED Group | Prospective TED/NTT Group | Prospective TED/TED Group
Started | 24 | 5 | 0 | 0
Completed | 20 | 4 | 0 | 0
Not Completed | 4 | 1 | 0 | 0
Not completed — Inform consent not signed by participant | 4 | 1 | 0 | 0
Period: Prospective Period
Arm/Group | Retrospective TED/NTT Group | Retrospective TED/TED Group | Prospective TED/NTT Group | Prospective TED/TED Group
Started | 0 | 0 | 5 (Participants were enrolled from retrospective period.) | 19 (Participants were enrolled from retrospective period.)
Completed | 0 | 0 | 4 | 15
Not Completed | 0 | 0 | 1 | 4
Not completed — Discontinued the study early but didn't complete an ET Visit. | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: Safety population included all enrolled participants who provided informed consent for the prospective portion and met all the inclusion criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Retrospective TED/NTT Group | Retrospective TED/TED Group | Total
Number analyzed (Participants) | 24 | 5 | 29
Age, Continuous [Mean (Standard Deviation); unit: Years] | 4.0 (2.88) | 8.2 (5.50) | 4.7 (3.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 0 | 9
  Male | 15 | 5 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 9 | 1 | 10
  Ethnicity: Not Hispanic or Latino | 15 | 3 | 18
  Ethnicity: Not allowed based on local regulations | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 20 | 3 | 23
  Race: Black or African American | 2 | 1 | 3
  Race: Asian | 0 | 1 | 1
  Race: Other | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) in Retrospective Observation Period
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. A SAE was any untoward medical occurrence (whether considered to be related to investigational product or not) that at any dose: results in death, was life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, was a congenital abnormality/birth defect, was an important medical event. Number of participants with AEs, related AEs, serious adverse events (SAEs) and related SAEs of retrospective observation period were reported.
Time Frame: From end of the core study (TED-C13-003 [NCT01952080]) up to the beginning of the prospective period (up to Week 168)
Population: Retrospective participants (RETRO): all participants who consented to participation in this extension study and provided data for the retrospective period of the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Retrospective TED/NTT Group | Retrospective TED/TED Group
Number analyzed (Participants) | 24 | 5
Participants
  Participants with AEs | 23 | 4
  Participants with Related AEs | 23 | 4
  Participants with SAEs | 23 | 4
  Participants with Related SAE | 0 | 0

2. Primary Outcome: Change From Baseline in Height for Age Z-score up to Week 168 of Retrospective Observation Period
Description: Height was measured using age Z-score. Z-score was calculated as (observed value - median value of the reference population) / standard deviation value of reference population. Centers for Disease Control and Prevention (age greater than or equal to [>=] 2 years old) and World Health Organization (age less than [<] 2 years old) Z-score calculation charts are used for calculation. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in height for age Z-score up to Week 168 of retrospective observation period was reported. Data for this outcome was not planned to be collected and analyzed in retrospective TED/TED group.
Time Frame: Baseline (Baseline visit in the core study [TED-C13-003 (NCT01952080)]) up to the beginning of the prospective period (up to Week 168)
Population: RETRO participants: all participants who consented to participation in this extension study and provided data for the retrospective period of the protocol. Here, overall number of participants analyzed signifies participants who were evaluable for this outcome measure. Data were not planned to be collected and analyzed for the retrospective TED/TED group.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Retrospective TED/NTT Group
Number analyzed (Participants) | 2
Z-score | 0.128 (0.0505)

3. Primary Outcome: Change From Baseline in Body Weight for Age Z-score up to Week 168 of Retrospective Observation Period
Description: Body weight was measured using age Z-score. Z-score was calculated as (observed value - median value of the reference population) / standard deviation value of reference population. Centers for Disease Control and Prevention (age >= 2 years old) and World Health Organization (age < 2 years old) Z-score calculation charts are used for calculation. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in body weight for age Z-score up to Week 168 was reported. Data for this outcome was not planned to be collected and analyzed in retrospective TED/TED group.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Retrospective TED/NTT Group
Number analyzed (Participants) | 2
Z-score | -0.181 (0.0601)

4. Primary Outcome: Change From Baseline in Body Mass Index (BMI) for Age Z-score up to Week 168 of Retrospective Observation Period
Description: BMI Z-score was calculated by using the retrospective height and weight data. Z-score was calculated as (observed value - median value of the reference population) / standard deviation value of reference population. Centers for Disease Control and Prevention (age >= 2 years old) and World Health Organization (age < 2 years old) Z-score calculation charts are used for calculation. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in height for age Z-score up to Week 168 of retrospective observation period was reported. Data for this outcome was not planned to be collected and analyzed in retrospective TED/TED group.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Retrospective TED/NTT Group
Number analyzed (Participants) | 2
Z-score | -0.283 (0.0646)

5. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) of Prospective Study Period
Description: TEAEs are defined as AEs that started or worsened on or after the first dose of teduglutide treatment in the core study. A SAE was any untoward medical occurrence (whether considered to be related to investigational product or not) that at any dose: results in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, was a congenital abnormality/birth defect, was an important medical event. AESI was an TEAE or TESAE of scientific and medical concern specific to the sponsor's product or program and for which ongoing monitoring and immediate notification by the investigator to the sponsor. Number of participants With TEAEs, treatment -emergent serious adverse events (TESAEs) and adverse events of special interest (AESI) of Prospective study period were reported.
Time Frame: From the beginning of the prospective study period to End of Study (EOS) (up to Week 144)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Prospective TED/NTT Group | Prospective TED/TED Group
Number analyzed (Participants) | 5 | 19
Participants
  Participants with TEAEs | 4 | 19
  Participants with TESAEs | 3 | 17
  Participants with AESI | 0 | 0

6. Primary Outcome: Change From Baseline in Height for Age Z-score up to Cycle 6 Week 12 During the End of Teduglutide Treatment Period of Prospective Study Period
Description: Height was measured using age Z-score. Z-score was calculated as (observed value - median value of the reference population) / standard deviation value of reference population. Centers for Disease Control and Prevention (age >= 2 years old) and World Health Organization (age < 2 years old) Z-score calculation charts are used for calculation. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in height for age Z-score up to Cycle 6 Week 12 during the end of teduglutide treatment period in prospective study period was reported.
Time Frame: Baseline (from the beginning of the prospective study period) up to Cycle 6 Week 12
Population: Safety population included all enrolled participants who provided informed consent for the prospective portion and met all the inclusion criteria. Here, overall number of participants analyzed signifies participants who were evaluable for this outcome measure. Data were not planned to be collected and analyzed for the prospective TED/NTT group.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Prospective TED/TED Group
Number analyzed (Participants) | 3
Z-score | 0.05 (1.068)

7. Primary Outcome: Change From Baseline in Body Weight for Age Z-score up to Cycle 6 Week 24 During the End of Teduglutide Treatment Period of Prospective Study Period
Description: Body weight was measured using age Z-score. Z-score was calculated as (observed value - median value of the reference population) / standard deviation value of reference population. Centers for Disease Control and Prevention (age >= 2 years old) and World Health Organization (age < 2 years old) Z-score calculation charts are used for calculation. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in body weight for age Z-score up to Cycle 6 Week 24 during the end of teduglutide treatment period of prospective study period was reported.
Time Frame: Baseline (from the beginning of the prospective study period) up to Cycle 6 Week 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Prospective TED/TED Group
Number analyzed (Participants) | 1
Z-score | -0.66 (NA) — Standard deviation could not be calculated because single participant was analyzed.

8. Primary Outcome: Change From Baseline in BMI for Age Z-score up to Cycle 6 Week 12 During the End of Teduglutide Treatment Period of Prospective Study Period
Description: BMI Z-score was calculated by using the height and weight data. Z-score was calculated as (observed value - median value of the reference population) / standard deviation value of reference population. Centers for Disease Control and Prevention (age >= 2 years old) and World Health Organization (age < 2 years old) Z-score calculation charts are used for calculation. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in BMI for age Z-score up to Cycle 6 Week 12 during the end of teduglutide treatment period of prospective study period was reported.
Time Frame: Baseline (from the beginning of the prospective study period) up to Cycle 6 Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Prospective TED/TED Group
Number analyzed (Participants) | 3
Z-score | -0.68 (0.349)

9. Primary Outcome: Average Total 48-Hour Urine Output up to Cycle 6 Week 12 During the End of Teduglutide Treatment Period of Prospective Study Period
Description: Average total urine output was calculated based on the daily data recorded in participants diaries over a 48-hour period of nutritional stability prior to each scheduled visit. Average total 48-Hour urine output up to Cycle 6 Week 12 during the end of teduglutide treatment period of prospective study period was reported. Here, mL/kg/day is abbreviated as milliliter per kilogram per day.
Time Frame: Baseline (from the beginning of the prospective study period) up to Cycle 6 Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mL/kg/day
Arm/Group | Prospective TED/TED Group
Number analyzed (Participants) | 3
mL/kg/day | 14.38 (12.712)

10. Primary Outcome: Average Total 48-Hour Urine Output up to Week 108 During the End of Non-Teduglutide Treatment (NTT) Period of Prospective Study Period
Description: Average total urine output was calculated based on the daily data recorded in participants diaries over a 48-hour period of nutritional stability prior to each scheduled visit. Average total 48-Hour urine output up to Week 108 during the end of NTT period in prospective study period was reported.
Time Frame: Baseline (from the beginning of the prospective study period) up to Week 108
Population: Safety population included all enrolled participants who provided informed consent for the prospective portion and met all the inclusion criteria. Here, overall number of participants analyzed signifies participants who were evaluable for this outcome measure. Data were not planned to be collected and analyzed for the prospective TED/TED group.
Measure: Mean (Standard Deviation); unit: mL/kg/day
Arm/Group | Prospective TED/NTT Group
Number analyzed (Participants) | 2
mL/kg/day | 22.86 (9.956)

11. Primary Outcome: Average Number of Stools Per Day up to Cycle 6 Week 24 During the End of Teduglutide Treatment Period of Prospective Study Period
Description: Average number of stools per day was calculated based on the daily data recorded in participants diaries over a 48-hour period of nutritional stability prior to each scheduled visit. Average number of stools per day up to cycle 6 week 24 during the end of teduglutide treatment period in prospective study period was reported.
Time Frame: Baseline (from the beginning of the prospective study period) up to Cycle 6 Week 24
Population: Safety population included all enrolled participants who provided informed consent for the prospective portion and met all the inclusion criteria. Here, overall number of participants analyzed signifies participants who were evaluable for this outcome measure. Data for this outcome was not planned to be collected and analyzed in prospective TED/NTT group.
Measure: Mean (Standard Deviation); unit: Stools per day
Arm/Group | Prospective TED/TED Group
Number analyzed (Participants) | 1
Stools per day | 5.50 (NA) — Standard deviation could not be calculated because single participant was analyzed.

12. Primary Outcome: Average Number of Stools Per Day up to Week 120 During the End of NTT Period of Prospective Study Period
Description: Average number of stools per day was calculated based on the daily data recorded in participants diaries over a 48-hour period of nutritional stability prior to each scheduled visit. Average number of stools per day up to Week 120 during the end of NTT period in prospective study period was reported.
Time Frame: Baseline (from the beginning of the prospective study period) up to Week 120
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Stools per day
Arm/Group | Prospective TED/NTT Group
Number analyzed (Participants) | 2
Stools per day | 3.75 (3.182)

13. Primary Outcome: Number of Participants With Positive Specific Antibodies at EOS During the End of Teduglutide Treatment Period of Prospective Study Period
Description: Number of participants with positive specific antibodies to teduglutide were used to summarize the presence of antibodies.
Time Frame: From the beginning of the prospective study period, EOS (up to Week 156)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Prospective TED/TED Group
Number analyzed (Participants) | 7
Participants | 1

14. Secondary Outcome: Number of Participants Achieved At Least 20 Percent (%) Reduction in Parenteral Support (PS) Volume at 12 Weeks Interval up to Week 156 of Retrospective Observation Period
Description: Number of participants achieved at least 20% reduction in PS volume at 12 weeks interval up to Week 156 in retrospective observation period was reported.
Time Frame: At Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, and 156
Population: RETRO participants: all participants who consented to participation in this extension study and provided data for the retrospective period of the protocol. Here, number analyzed signifies participants who were evaluable for this outcome at specific time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Retrospective TED/NTT Group | Retrospective TED/TED Group
Number analyzed (Participants) | 24 | 5
Participants
  At Week 12 | 12 | 2
  At Week 24: number analyzed (Participants) | 23 | 5
  At Week 24 | 9 | 2
  At Week 36: number analyzed (Participants) | 24 | 4
  At Week 36 | 9 | 4
  At Week 48: number analyzed (Participants) | 23 | 4
  At Week 48 | 9 | 4
  At Week 60: number analyzed (Participants) | 23 | 5
  At Week 60 | 9 | 4
  At Week 72: number analyzed (Participants) | 22 | 5
  At Week 72 | 6 | 2
  At Week 84: number analyzed (Participants) | 22 | 5
  At Week 84 | 7 | 2
  At Week 96 | 10 | 5
  At Week 108 | 9 | 5
  At Week 120: number analyzed (Participants) | 22 | 5
  At Week 120 | 10 | 4
  At Week 132: number analyzed (Participants) | 14 | 4
  At Week 132 | 7 | 4
  At Week 144: number analyzed (Participants) | 8 | 1
  At Week 144 | 3 | 1
  At Week 156: number analyzed (Participants) | 2 | 1
  At Week 156 | 0 | 1

15. Secondary Outcome: Change From Baseline in PS Volume at 12 Weeks Interval up to Week 156 of Retrospective Observation Period
Description: Change from baseline in PS volume at 12 weeks interval up to Week 156 in retrospective observation period was reported.
Time Frame: Baseline (Baseline visit in the core study [TED-C13-003 (NCT01952080)]), Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, and 156
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mL/kg/day
Arm/Group | Retrospective TED/NTT Group | Retrospective TED/TED Group
Number analyzed (Participants) | 24 | 5
mL/kg/day
  Change at Week 12: number analyzed (Participants) | 23 | 5
  Change at Week 12 | -14.45 (17.770) | -12.84 (17.694)
  Change at Week 24 | -9.27 (21.642) | -13.49 (14.530)
  Change at Week 36: number analyzed (Participants) | 23 | 5
  Change at Week 36 | -10.65 (20.877) | -17.91 (17.069)
  Change at Week 48: number analyzed (Participants) | 23 | 4
  Change at Week 48 | -12.24 (29.646) | -26.12 (8.044)
  Change at Week 60: number analyzed (Participants) | 23 | 5
  Change at Week 60 | -13.85 (30.219) | -21.35 (12.285)
  Change at Week 72: number analyzed (Participants) | 22 | 5
  Change at Week 72 | -13.65 (30.577) | -11.41 (22.030)
  Change at Week 84: number analyzed (Participants) | 22 | 5
  Change at Week 84 | -8.74 (36.078) | -15.65 (19.603)
  Change at Week 96 | -12.87 (37.996) | -27.34 (16.531)
  Change at Week 108 | -10.35 (29.370) | -31.83 (14.872)
  Change at Week 120: number analyzed (Participants) | 22 | 5
  Change at Week 120 | -12.21 (27.480) | -30.48 (19.043)
  Change at Week 132: number analyzed (Participants) | 14 | 4
  Change at Week 132 | -19.20 (26.171) | -37.70 (12.296)
  Change at Week 144: number analyzed (Participants) | 8 | 1
  Change at Week 144 | -16.79 (29.620) | -34.32 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Change at Week 156: number analyzed (Participants) | 2 | 1
  Change at Week 156 | -7.46 (1.931) | -34.43 (NA) — Standard deviation could not be calculated because single participant was analyzed.

16. Secondary Outcome: Percent Change From Baseline in PS Volume at 12 Weeks Interval up to Week 156 of Retrospective Observation Period
Description: Percent change from baseline in PS volume at 12 weeks interval up to Week 156 of retrospective observation period was reported.
Time Frame: as for outcome 15
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Retrospective TED/NTT Group | Retrospective TED/TED Group
Number analyzed (Participants) | 24 | 5
Percent change
  Percent change at Week 12: number analyzed (Participants) | 23 | 5
  Percent change at Week 12 | -24.50 (27.853) | -24.88 (35.649)
  Percent change at Week 24: number analyzed (Participants) | 24 | 4
  Percent change at Week 24 | -10.72 (33.081) | -32.10 (31.645)
  Percent change at Week 36: number analyzed (Participants) | 23 | 5
  Percent change at Week 36 | -13.21 (34.172) | -43.09 (42.753)
  Percent change at Week 48: number analyzed (Participants) | 23 | 4
  Percent change at Week 48 | -14.04 (39.390) | -65.18 (31.650)
  Percent change at Week 60: number analyzed (Participants) | 23 | 5
  Percent change at Week 60 | -16.15 (39.491) | -53.61 (37.141)
  Percent change at Week 72: number analyzed (Participants) | 22 | 5
  Percent change at Week 72 | -14.19 (40.558) | -14.11 (58.452)
  Percent change at Week 84: number analyzed (Participants) | 22 | 5
  Percent change at Week 84 | -8.67 (47.108) | -30.25 (39.598)
  Percent change at Week 96 | -12.04 (51.631) | -61.19 (29.335)
  Percent change at Week 108 | -10.62 (48.820) | -73.43 (29.298)
  Percent change at Week 120: number analyzed (Participants) | 22 | 5
  Percent change at Week 120 | -12.89 (49.366) | -69.61 (39.194)
  Percent change at Week 132: number analyzed (Participants) | 14 | 4
  Percent change at Week 132 | -20.24 (47.431) | -85.92 (17.457)
  Percent change at Week 144: number analyzed (Participants) | 8 | 1
  Percent change at Week 144 | -7.70 (44.170) | -65.20 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Percent change at Week 156: number analyzed (Participants) | 2 | 1
  Percent change at Week 156 | -17.21 (3.164) | -65.42 (NA) — Standard deviation could not be calculated because single participant was analyzed.

17. Secondary Outcome: Change From Baseline in PS Caloric Intake at 12 Weeks Interval up to Week 156 of Retrospective Observation Period
Description: Change from baseline in PS caloric intake at 12 weeks interval up to Week 156 of retrospective observation period was reported. Here, kilo-calories per kilogram per day was abbreviated as (kcal/kg/day).
Time Frame: as for outcome 15
Population: RETRO participants: all participants who consented to participation in this extension study and provided data for the retrospective period of the protocol. Here, overall number of participants analyzed signifies participants who were evaluable for this outcome and number analyzed signifies participants who were evaluable at specific time point.
Measure: Mean (Standard Deviation); unit: kcal/kg/day
Arm/Group | Retrospective TED/NTT Group | Retrospective TED/TED Group
Number analyzed (Participants) | 23 | 5
kcal/kg/day
  Change at Week 12 | -10.15 (13.026) | -2.64 (18.739)
  Change at Week 24: number analyzed (Participants) | 23 | 4
  Change at Week 24 | -3.96 (16.970) | -7.25 (11.916)
  Change at Week 36: number analyzed (Participants) | 22 | 5
  Change at Week 36 | -8.38 (17.148) | -6.42 (24.547)
  Change at Week 48: number analyzed (Participants) | 22 | 4
  Change at Week 48 | -9.84 (22.144) | -18.11 (7.896)
  Change at Week 60: number analyzed (Participants) | 22 | 5
  Change at Week 60 | -10.55 (23.136) | -10.53 (18.538)
  Change at Week 72: number analyzed (Participants) | 21 | 5
  Change at Week 72 | -12.64 (23.642) | -0.05 (23.552)
  Change at Week 84: number analyzed (Participants) | 21 | 5
  Change at Week 84 | -9.70 (24.860) | -5.24 (23.064)
  Change at Week 96 | -10.08 (23.998) | -15.09 (18.604)
  Change at Week 108 | -7.20 (22.875) | -19.05 (18.229)
  Change at Week 120: number analyzed (Participants) | 21 | 5
  Change at Week 120 | -7.98 (21.425) | -17.18 (23.169)
  Change at Week 132: number analyzed (Participants) | 13 | 4
  Change at Week 132 | -12.93 (18.744) | -27.59 (5.114)
  Change at Week 144: number analyzed (Participants) | 8 | 1
  Change at Week 144 | -11.97 (17.977) | -25.53 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Change at Week 156: number analyzed (Participants) | 2 | 1
  Change at Week 156 | -6.55 (4.708) | -25.67 (NA) — Standard deviation could not be calculated because single participant was analyzed.

18. Secondary Outcome: Percent Change From Baseline in PS Caloric Intake at 12 Weeks Interval up to Week 156 of Retrospective Observation Period
Description: Percent change from baseline in PS caloric intake at 12 weeks interval up to Week 156 of retrospective observation period was reported.
Time Frame: as for outcome 15
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Retrospective TED/NTT Group | Retrospective TED/TED Group
Number analyzed (Participants) | 23 | 5
Percent change
  Percent change at Week 12 | -24.91 (29.001) | 7.64 (82.061)
  Percent change at Week 24: number analyzed (Participants) | 23 | 4
  Percent change at Week 24 | -10.12 (42.431) | -21.29 (37.759)
  Percent change at Week 36: number analyzed (Participants) | 22 | 5
  Percent change at Week 36 | -18.29 (41.070) | -3.38 (118.167)
  Percent change at Week 48: number analyzed (Participants) | 22 | 4
  Percent change at Week 48 | -21.03 (43.924) | -59.31 (38.042)
  Percent change at Week 60: number analyzed (Participants) | 22 | 5
  Percent change at Week 60 | -20.63 (44.903) | -25.65 (83.470)
  Percent change at Week 72: number analyzed (Participants) | 21 | 5
  Percent change at Week 72 | -25.48 (45.035) | 23.26 (99.380)
  Percent change at Week 84: number analyzed (Participants) | 21 | 5
  Percent change at Week 84 | -20.42 (45.287) | 4.41 (102.162)
  Percent change at Week 96 | -21.12 (46.005) | -36.49 (72.357)
  Percent change at Week 108 | -16.41 (46.034) | -50.24 (70.513)
  Percent change at Week 120: number analyzed (Participants) | 21 | 5
  Percent change at Week 120 | -18.79 (45.774) | -38.58 (97.750)
  Percent change at Week 132: number analyzed (Participants) | 13 | 4
  Percent change at Week 132 | -29.37 (40.170) | -82.01 (21.165)
  Percent change at Week 144: number analyzed (Participants) | 8 | 1
  Percent change at Week 144 | -25.25 (33.618) | -60.36 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Percent change at Week 156: number analyzed (Participants) | 2 | 1
  Percent change at Week 156 | -15.66 (7.700) | -60.69 (NA) — Standard deviation could not be calculated because single participant was analyzed.

19. Secondary Outcome: Change From Baseline in Number of Hours Per Day of PS Usage at 12 Weeks Interval up to Week 156 of Retrospective Observation Period
Description: Data for this outcome measure was not analyzed and collected because changes from baseline for prescribed hours per day were not collected at baseline in the core study.
Time Frame: Baseline (Baseline visit in the core study [TED-C13-003 (NCT01952080)]) up to Week 156
Population: Data for this outcome measure was not analyzed and collected because changes from baseline for prescribed hours per day were not collected at baseline in the core study.
Arm/Group | Retrospective TED/NTT Group | Retrospective TED/TED Group
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Percent Change From Baseline in Number of Hours Per Day of PS Usage at 12 Weeks Interval up to Week 156 of Retrospective Observation Period
Description: Data for this outcome measure was not analyzed and collected because changes from baseline for prescribed hours per day were not collected at baseline in the core study. Hence, percent change was not assessed in this study.
Time Frame: Baseline (Baseline visit in the core study [TED-C13-003 (NCT01952080)]) up to Week 156
Population: as for outcome 19
Arm/Group | Retrospective TED/NTT Group | Retrospective TED/TED Group
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Change From Baseline in Number of Days Per Week of PS Usage at 12 Weeks Interval up to Week 156 of Retrospective Observation Period
Description: Change from baseline in number of days per Week of PS usage at 12 weeks interval up to Week 156 in retrospective observation period was reported.
Time Frame: as for outcome 15
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Days per week
Arm/Group | Retrospective TED/NTT Group | Retrospective TED/TED Group
Number analyzed (Participants) | 24 | 5
Days per week
  Change at Week 12 | -0.38 (1.469) | -1.20 (2.683)
  Change at Week 24: number analyzed (Participants) | 24 | 4
  Change at Week 24 | -0.29 (1.429) | -1.00 (2.000)
  Change at Week 36: number analyzed (Participants) | 23 | 5
  Change at Week 36 | -0.43 (1.562) | -2.60 (2.793)
  Change at Week 48: number analyzed (Participants) | 23 | 4
  Change at Week 48 | -0.61 (2.017) | -4.50 (2.082)
  Change at Week 60: number analyzed (Participants) | 23 | 5
  Change at Week 60 | -0.61 (2.017) | -3.00 (3.536)
  Change at Week 72: number analyzed (Participants) | 22 | 5
  Change at Week 72 | -0.64 (2.060) | -1.40 (2.966)
  Change at Week 84: number analyzed (Participants) | 22 | 5
  Change at Week 84 | -0.64 (2.060) | -1.40 (2.966)
  Change at Week 96 | -1.17 (2.665) | -2.00 (3.536)
  Change at Week 108 | -0.88 (2.365) | -3.80 (3.701)
  Change at Week 120: number analyzed (Participants) | 22 | 5
  Change at Week 120 | -0.95 (2.459) | -3.80 (3.701)
  Change at Week 132: number analyzed (Participants) | 14 | 4
  Change at Week 132 | -1.00 (2.542) | -5.25 (2.062)
  Change at Week 144: number analyzed (Participants) | 8 | 1
  Change at Week 144 | 0.00 (0.000) | -3.00 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Change at Week 156: number analyzed (Participants) | 2 | 1
  Change at Week 156 | 0.00 (0.000) | -3.00 (NA) — Standard deviation could not be calculated because single participant was analyzed.

22. Secondary Outcome: Percent Change From Baseline in Number of Days Per Week of PS Usage at 12 Weeks Interval up to Week 156 of Retrospective Observation Period
Description: Percent change from baseline in number of days per Week of PS usage at 12 weeks interval up to Week 156 in retrospective observation period was reported.
Time Frame: as for outcome 15
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Retrospective TED/NTT Group | Retrospective TED/TED Group
Number analyzed (Participants) | 24 | 5
Percent change
  Percent change at Week 12 | -6.25 (22.421) | -14.86 (41.913)
  Percent change at Week 24: number analyzed (Participants) | 24 | 4
  Percent change at Week 24 | -4.17 (20.412) | -14.29 (28.571)
  Percent change at Week 36: number analyzed (Participants) | 23 | 5
  Percent change at Week 36 | -6.21 (22.309) | -34.86 (44.648)
  Percent change at Week 48: number analyzed (Participants) | 23 | 4
  Percent change at Week 48 | -8.70 (28.810) | -64.29 (29.738)
  Percent change at Week 60: number analyzed (Participants) | 23 | 5
  Percent change at Week 60 | -8.70 (28.810) | -40.57 (54.638)
  Percent change at Week 72: number analyzed (Participants) | 22 | 5
  Percent change at Week 72 | -9.09 (29.424) | -17.71 (45.821)
  Percent change at Week 84: number analyzed (Participants) | 22 | 5
  Percent change at Week 84 | -9.09 (29.424) | -17.71 (45.821)
  Percent change at Week 96 | -16.67 (38.069) | -26.29 (53.886)
  Percent change at Week 108 | -12.50 (33.783) | -52.00 (57.407)
  Percent change at Week 120: number analyzed (Participants) | 22 | 5
  Percent change at Week 120 | -13.64 (35.125) | -52.00 (57.407)
  Percent change at Week 132: number analyzed (Participants) | 14 | 4
  Percent change at Week 132 | -14.29 (36.314) | -75.00 (29.451)
  Percent change at Week 144: number analyzed (Participants) | 8 | 1
  Percent change at Week 144 | 0.00 (0.000) | -42.86 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Percent change at Week 156: number analyzed (Participants) | 2 | 1
  Percent change at Week 156 | 0.00 (0.000) | -42.86 (NA) — Standard deviation could not be calculated because single participant was analyzed.

23. Secondary Outcome: Number of Participants Who Achieved At Least 20, 50 and 75% Reduction in PS Volume at EOT of Each Cycle During the End of Teduglutide Treatment Period of Prospective Study Period
Description: Number of participants who achieved at least 20, 50 and 75% reduction in PS volume at EOT of each cycle during the end of teduglutide treatment period in prospective study period was reported.
Time Frame: At EOT of each Cycles 1 to 6 (up to Week 140) (length of each Cycle 1 to 5 = 24 weeks, length of Cycle 6 = 20 weeks)
Population: Safety population included all enrolled participants who provided informed consent for the prospective portion and met all the inclusion criteria. Here, number analyzed signifies participants who were evaluable for this outcome at specific time point. Data were not planned to be collected and analyzed for the prospective TED/NTT group.
Measure: Count of Participants; unit: Participants
Arm/Group | Prospective TED/TED Group
Number analyzed (Participants) | 19
Participants
  Cycle 1: EOT at >= 20% | 13
  Cycle 2: EOT at >= 20%: number analyzed (Participants) | 17
  Cycle 2: EOT at >= 20% | 12
  Cycle 3: EOT at >= 20%: number analyzed (Participants) | 14
  Cycle 3: EOT at >= 20% | 10
  Cycle 4: EOT at >= 20%: number analyzed (Participants) | 13
  Cycle 4: EOT at >= 20% | 9
  Cycle 5: EOT at >= 20%: number analyzed (Participants) | 8
  Cycle 5: EOT at >= 20% | 7
  Cycle 6: EOT at >= 20%: number analyzed (Participants) | 5
  Cycle 6: EOT at >= 20% | 5
  Cycle 1: EOT at >= 50% | 5
  Cycle 2: EOT at >= 50%: number analyzed (Participants) | 17
  Cycle 2: EOT at >= 50% | 10
  Cycle 3: EOT at >= 50%: number analyzed (Participants) | 14
  Cycle 3: EOT at >= 50% | 9
  Cycle 4: EOT at >= 50%: number analyzed (Participants) | 13
  Cycle 4: EOT at >= 50% | 9
  Cycle 5: EOT at >= 50%: number analyzed (Participants) | 8
  Cycle 5: EOT at >= 50% | 5
  Cycle 6: EOT at >= 50%: number analyzed (Participants) | 5
  Cycle 6: EOT at >= 50% | 4
  Cycle 1: EOT at >= 75% | 2
  Cycle 2: EOT at >= 75%: number analyzed (Participants) | 17
  Cycle 2: EOT at >= 75% | 4
  Cycle 3: EOT at >= 75%: number analyzed (Participants) | 14
  Cycle 3: EOT at >= 75% | 6
  Cycle 4: EOT at >= 75%: number analyzed (Participants) | 13
  Cycle 4: EOT at >= 75% | 5
  Cycle 5: EOT at >= 75%: number analyzed (Participants) | 8
  Cycle 5: EOT at >= 75% | 4
  Cycle 6: EOT at >= 75%: number analyzed (Participants) | 5
  Cycle 6: EOT at >= 75% | 3

24. Secondary Outcome: Change From Baseline in PS Volume at EOT of Each Cycle During the End of Teduglutide Treatment Period of Prospective Study Period
Description: Change from baseline in PS volume at EOT of each cycle during the end of teduglutide treatment period in prospective study period was reported.
Time Frame: Baseline (from the beginning of the prospective study period), EOT of each Cycles 1 to 6 (up to Week 136) (length of each Cycle 1 to 5 = 24 weeks, length of Cycle 6 = 16 weeks)
Population: Safety population included all enrolled participants who provided informed consent for the prospective portion and met all the inclusion criteria. Here, overall number of participants analyzed signifies participants who were evaluable for this outcome measure and number analyzed signifies participants who were evaluable at specific time point. Data were not planned to be collected and analyzed for the prospective TED/NTT group.
Measure: Mean (Standard Deviation); unit: mL/kg/day
Arm/Group | Prospective TED/TED Group
Number analyzed (Participants) | 18
mL/kg/day
  Change at Cycle 1: EOT | -25.18 (19.915)
  Change at Cycle 2: EOT: number analyzed (Participants) | 16
  Change at Cycle 2: EOT | -28.59 (29.856)
  Change at Cycle 3: EOT: number analyzed (Participants) | 13
  Change at Cycle 3: EOT | -40.05 (29.711)
  Change at Cycle 4: EOT: number analyzed (Participants) | 12
  Change at Cycle 4: EOT | -40.10 (30.359)
  Change at Cycle 5: EOT: number analyzed (Participants) | 7
  Change at Cycle 5: EOT | -40.49 (24.259)
  Change at Cycle 6: EOT: number analyzed (Participants) | 5
  Change at Cycle 6: EOT | -47.57 (26.243)

25. Secondary Outcome: Percent Change From Baseline in PS Volume at EOT of Each Cycle During the End of Teduglutide Treatment Period of Prospective Study Period
Description: Percent change from baseline in PS volume at EOT of each cycle during the end of teduglutide treatment period in prospective study period.
Time Frame: as for outcome 24
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Prospective TED/TED Group
Number analyzed (Participants) | 18
Percent change
  Percent change: Cycle 1: EOT | -38.02 (28.611)
  Percent change: Cycle 2: EOT: number analyzed (Participants) | 16
  Percent change: Cycle 2: EOT | -45.58 (48.150)
  Percent change: Cycle 3: EOT: number analyzed (Participants) | 13
  Percent change: Cycle 3: EOT | -62.16 (41.805)
  Percent change: Cycle 4: EOT: number analyzed (Participants) | 12
  Percent change: Cycle 4: EOT | -62.92 (38.466)
  Percent change: Cycle 5: EOT: number analyzed (Participants) | 7
  Percent change: Cycle 5: EOT | -73.49 (34.593)
  Percent change: Cycle 6: EOT: number analyzed (Participants) | 5
  Percent change: Cycle 6: EOT | -78.75 (33.949)

26. Secondary Outcome: Change From Baseline in PS Caloric Intake at EOT of Each Cycle During the End of Teduglutide Treatment Period of Prospective Study Period
Description: Change from baseline in PS caloric intake at EOT of each cycle during the end of teduglutide treatment period in prospective study period was reported.
Time Frame: as for outcome 24
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: kcal/kg/day
Arm/Group | Prospective TED/TED Group
Number analyzed (Participants) | 19
kcal/kg/day
  Change at Cycle 1: EOT | -17.66 (17.649)
  Change at Cycle 2: EOT: number analyzed (Participants) | 17
  Change at Cycle 2: EOT | -19.95 (23.402)
  Change at Cycle 3: EOT: number analyzed (Participants) | 14
  Change at Cycle 3: EOT | -27.66 (19.668)
  Change at Cycle 4: EOT: number analyzed (Participants) | 13
  Change at Cycle 4: EOT | -24.05 (22.746)
  Change at Cycle 5: EOT: number analyzed (Participants) | 8
  Change at Cycle 5: EOT | -26.98 (27.465)
  Change at Cycle 6: EOT: number analyzed (Participants) | 5
  Change at Cycle 6: EOT | -27.53 (32.486)

27. Secondary Outcome: Percent Change From Baseline in PS Caloric Intake at EOT of Each Cycle During the End of Teduglutide Treatment Period of Prospective Study Period
Description: Percent change from baseline in PS caloric intake at EOT of each cycle during the end of teduglutide treatment period in prospective study period was reported.
Time Frame: as for outcome 24
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Prospective TED/TED Group
Number analyzed (Participants) | 19
Percent change
  Percent change at Cycle 1: EOT | -33.50 (40.439)
  Percent change at Cycle 2: EOT: number analyzed (Participants) | 17
  Percent change at Cycle 2: EOT | -42.06 (44.077)
  Percent change at Cycle 3: EOT: number analyzed (Participants) | 14
  Percent change at Cycle 3: EOT | -62.47 (37.677)
  Percent change at Cycle 4: EOT: number analyzed (Participants) | 13
  Percent change at Cycle 4: EOT | -49.51 (54.041)
  Percent change at Cycle 5: EOT: number analyzed (Participants) | 8
  Percent change at Cycle 5: EOT | -54.08 (64.002)
  Percent change at Cycle 6: EOT: number analyzed (Participants) | 5
  Percent change at Cycle 6: EOT | -59.00 (57.267)

28. Secondary Outcome: Number of Participants Who Achieved 100% Reduction in Complete Weaning of PS Volume at EOT of Each Cycle During the End of Teduglutide Treatment Period of Prospective Study Period
Description: Number of participants who achieved at least 100% reduction in complete weaning of PS volume at EOT of each cycle during the end of teduglutide treatment period in prospective study period was reported.
Time Frame: At EOT of each Cycles 1 to 6 (up to Week 144) (length of each Cycle 1 to 6 = 24 weeks)
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Prospective TED/TED Group
Number analyzed (Participants) | 19
Participants
  Cycle 1: EOT | 1
  Cycle 2: EOT: number analyzed (Participants) | 17
  Cycle 2: EOT | 3
  Cycle 3: EOT: number analyzed (Participants) | 14
  Cycle 3: EOT | 6
  Cycle 4: EOT: number analyzed (Participants) | 13
  Cycle 4: EOT | 5
  Cycle 5: EOT: number analyzed (Participants) | 8
  Cycle 5: EOT | 4
  Cycle 6: EOT: number analyzed (Participants) | 5
  Cycle 6: EOT | 3

29. Secondary Outcome: Change From Baseline in Number of Hours Per Day of PS Usage at EOT of Each Cycle During the End of Teduglutide Treatment Period of Prospective Study Period
Description: Change from baseline in number of hours per day of PS usage at EOT of each cycle during the end of teduglutide treatment period in prospective study period was reported.
Time Frame: as for outcome 24
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Hours per day
Arm/Group | Prospective TED/TED Group
Number analyzed (Participants) | 18
Hours per day
  Change at Cycle 1: EOT | -3.40 (3.752)
  Change at Cycle 2: EOT: number analyzed (Participants) | 16
  Change at Cycle 2: EOT | -4.80 (5.360)
  Change at Cycle 3: EOT: number analyzed (Participants) | 13
  Change at Cycle 3: EOT | -6.69 (4.247)
  Change at Cycle 4: EOT: number analyzed (Participants) | 12
  Change at Cycle 4: EOT | -6.48 (4.881)
  Change at Cycle 5: EOT: number analyzed (Participants) | 7
  Change at Cycle 5: EOT | -6.71 (6.175)
  Change at Cycle 6: EOT: number analyzed (Participants) | 5
  Change at Cycle 6: EOT | -8.08 (6.075)

30. Secondary Outcome: Percent Change From Baseline in Number of Hours Per Day of PS Usage at EOT of Each Cycle During the End of Teduglutide Treatment Period of Prospective Study Period
Description: Percent change from baseline in number of hours per day of PS usage at EOT of each cycle during the end of teduglutide treatment period in prospective study period was reported.
Time Frame: as for outcome 24
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Prospective TED/TED Group
Number analyzed (Participants) | 18
Percent change
  Percent change at Cycle 1: EOT | -26.32 (29.732)
  Percent change at Cycle 2: EOT: number analyzed (Participants) | 16
  Percent change at Cycle 2: EOT | -40.47 (40.476)
  Percent change at Cycle 3: EOT: number analyzed (Participants) | 13
  Percent change at Cycle 3: EOT | -57.61 (36.973)
  Percent change at Cycle 4: EOT: number analyzed (Participants) | 12
  Percent change at Cycle 4: EOT | -55.87 (42.693)
  Percent change at Cycle 5: EOT: number analyzed (Participants) | 7
  Percent change at Cycle 5: EOT | -58.85 (52.717)
  Percent change at Cycle 6: EOT: number analyzed (Participants) | 5
  Percent change at Cycle 6: EOT | -66.39 (46.042)

31. Secondary Outcome: Change From Baseline in Number of Days Per Week of PS Usage at EOT of Each Cycle During the End of Teduglutide Treatment Period of Prospective Study Period
Description: Change from baseline in number of days per week of PS usage at EOT of each cycle during the end of teduglutide treatment period in prospective study period was reported.
Time Frame: as for outcome 24
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Days per week
Arm/Group | Prospective TED/TED Group
Number analyzed (Participants) | 18
Days per week
  Change at Cycle 1: EOT | -0.60 (1.892)
  Change at Cycle 2: EOT: number analyzed (Participants) | 16
  Change at Cycle 2: EOT | -1.93 (2.840)
  Change at Cycle 3: EOT: number analyzed (Participants) | 13
  Change at Cycle 3: EOT | -3.03 (3.257)
  Change at Cycle 4: EOT: number analyzed (Participants) | 12
  Change at Cycle 4: EOT | -2.99 (3.610)
  Change at Cycle 5: EOT: number analyzed (Participants) | 7
  Change at Cycle 5: EOT | -3.83 (3.969)
  Change at Cycle 6: EOT: number analyzed (Participants) | 5
  Change at Cycle 6: EOT | -4.37 (3.618)

32. Secondary Outcome: Percent Change From Baseline in Number of Days Per Week of PS Usage at EOT of Each Cycle During the End of Teduglutide Treatment Period of Prospective Study Period
Description: Percent change from baseline in number of days per week of PS usage at EOT of each cycle during the end of teduglutide treatment period in prospective study period was reported.
Time Frame: as for outcome 24
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Prospective TED/TED Group
Number analyzed (Participants) | 18
Percent change
  Percent change at Cycle 1: EOT | -9.01 (27.472)
  Percent change at Cycle 2: EOT: number analyzed (Participants) | 16
  Percent change at Cycle 2: EOT | -29.24 (40.525)
  Percent change at Cycle 3: EOT: number analyzed (Participants) | 13
  Percent change at Cycle 3: EOT | -44.51 (47.929)
  Percent change at Cycle 4: EOT: number analyzed (Participants) | 12
  Percent change at Cycle 4: EOT | -42.38 (51.929)
  Percent change at Cycle 5: EOT: number analyzed (Participants) | 7
  Percent change at Cycle 5: EOT | -54.29 (57.404)
  Percent change at Cycle 6: EOT: number analyzed (Participants) | 5
  Percent change at Cycle 6: EOT | -62.86 (51.110)

33. Other Pre Specified Outcome: Change From Baseline In Pediatric Quality of Life Inventory (PedsQL) Generic Core Scale (GCS) Score at Week 12 and 24 of Each Treatment Cycle During the Teduglutide Treatment Periods of Prospective Study Period
Description: PedsQL GCS was used for quality of life assessment. It encompasses 4 dimensions of functioning (physical, emotional, social, school). Age groups are: Toddler (2-4 years), Young child (5-7 years), Child (8-12 years), and Teens (13-18 years). Depending on the participants age, the questionnaire may be completed by either the participant or the parent/caregiver as appropriate. For the Toddler group, the PedsQL GCS consisted of 21 items, using a 5-point Likert scale (0 to 4); for all other groups, the PedsQL GCS consisted of 23 items, with a 3-point Likert scale (0, 2, 4) for the young child, and a 5-point Likert scale for the child and teens groups. Scores are transformed on a scale from 0 to 100 where 0=100, 1=75, 2=50, 3=25, and 4=0. Higher scores indicate improved quality of life.
Time Frame: Baseline (from the beginning of the prospective study period), Week 12 and 24 of Cycles 1 to 6
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Prospective TED/TED Group
Number analyzed (Participants) | 15
Score on a scale
  Physical Functioning: Change at Cycle 1 Week 12 | -0.39 (24.326)
  Physical Functioning: Change at Cycle 1 Week 24 | -0.83 (10.726)
  Physical Functioning: Change at Cycle 2 Week 12: number analyzed (Participants) | 12
  Physical Functioning: Change at Cycle 2 Week 12 | 2.34 (15.717)
  Physical Functioning: Change at Cycle 2 Week 24: number analyzed (Participants) | 13
  Physical Functioning: Change at Cycle 2 Week 24 | 2.40 (16.296)
  Physical Functioning: Change at Cycle 3 Week 12: number analyzed (Participants) | 11
  Physical Functioning: Change at Cycle 3 Week 12 | -0.57 (16.167)
  Physical Functioning: Change at Cycle 3 Week 24: number analyzed (Participants) | 9
  Physical Functioning: Change at Cycle 3 Week 24 | -1.74 (25.963)
  Physical Functioning: Change at Cycle 4 Week 12: number analyzed (Participants) | 9
  Physical Functioning: Change at Cycle 4 Week 12 | -1.74 (22.378)
  Physical Functioning: Change at Cycle 4 Week 24: number analyzed (Participants) | 7
  Physical Functioning: Change at Cycle 4 Week 24 | 1.79 (19.998)
  Physical Functioning: Change at Cycle 5 Week 12: number analyzed (Participants) | 5
  Physical Functioning: Change at Cycle 5 Week 12 | -7.50 (19.961)
  Physical Functioning: Change at Cycle 5 Week 24: number analyzed (Participants) | 4
  Physical Functioning: Change at Cycle 5 Week 24 | -2.34 (14.292)
  Physical Functioning: Change at Cycle 6 Week 12: number analyzed (Participants) | 4
  Physical Functioning: Change at Cycle 6 Week 12 | -6.25 (22.244)
  Physical Functioning: Change at Cycle 6 Week 24: number analyzed (Participants) | 1
  Physical Functioning: Change at Cycle 6 Week 24 | 3.13 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Emotional Functioning: Change at Cycle 1 Week 12 | 4.17 (18.843)
  Emotional Functioning: Change at Cycle 1 Week 24 | -4.67 (24.511)
  Emotional Functioning: Change at Cycle 2 Week 12: number analyzed (Participants) | 12
  Emotional Functioning: Change at Cycle 2 Week 12 | -3.33 (28.591)
  Emotional Functioning: Change at Cycle 2 Week 24: number analyzed (Participants) | 13
  Emotional Functioning: Change at Cycle 2 Week 24 | -0.38 (21.454)
  Emotional Functioning: Change at Cycle 3 Week 12: number analyzed (Participants) | 11
  Emotional Functioning: Change at Cycle 3 Week 12 | 7.05 (29.661)
  Emotional Functioning: Change at Cycle 3 Week 24: number analyzed (Participants) | 9
  Emotional Functioning: Change at Cycle 3 Week 24 | -8.33 (36.120)
  Emotional Functioning: Change at Cycle 4 Week 12: number analyzed (Participants) | 9
  Emotional Functioning: Change at Cycle 4 Week 12 | 2.78 (33.481)
  Emotional Functioning: Change at Cycle 4 Week 24: number analyzed (Participants) | 7
  Emotional Functioning: Change at Cycle 4 Week 24 | -0.71 (35.786)
  Emotional Functioning: Change at Cycle 5 Week 12: number analyzed (Participants) | 5
  Emotional Functioning: Change at Cycle 5 Week 12 | -11.00 (40.566)
  Emotional Functioning: Cycle 5 Week 24: number analyzed (Participants) | 4
  Emotional Functioning: Cycle 5 Week 24 | -17.50 (37.804)
  Emotional Functioning: Change at Cycle 6 Week 12: number analyzed (Participants) | 4
  Emotional Functioning: Change at Cycle 6 Week 12 | -5.63 (56.065)
  Emotional Functioning: Change at Cycle 6 Week 24: number analyzed (Participants) | 1
  Emotional Functioning: Change at Cycle 6 Week 24 | 17.50 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Social Functioning: Change at Cycle 1 Week 12: number analyzed (Participants) | 1
  Social Functioning: Change at Cycle 1 Week 12 | -15.00 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Social Functioning: Change at Cycle 1 Week 24: number analyzed (Participants) | 1
  Social Functioning: Change at Cycle 1 Week 24 | -10.00 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Social Functioning: Change at Cycle 2 Week 12: number analyzed (Participants) | 1
  Social Functioning: Change at Cycle 2 Week 12 | -5.00 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Social Functioning: Change at Cycle 2 Week 24: number analyzed (Participants) | 1
  Social Functioning: Change at Cycle 2 Week 24 | 0.00 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Social Functioning: Change at Cycle 3 Week 12: number analyzed (Participants) | 1
  Social Functioning: Change at Cycle 3 Week 12 | 10.00 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Social Functioning: Change at Cycle 3 Week 24: number analyzed (Participants) | 1
  Social Functioning: Change at Cycle 3 Week 24 | 0.00 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Social Functioning: Change at Cycle 4 Week 12: number analyzed (Participants) | 1
  Social Functioning: Change at Cycle 4 Week 12 | 10.00 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Social Functioning: Change at Cycle 4 Week 24: number analyzed (Participants) | 1
  Social Functioning: Change at Cycle 4 Week 24 | 10.00 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Social Functioning: Change at Cycle 5 Week 12: number analyzed (Participants) | 1
  Social Functioning: Change at Cycle 5 Week 12 | 10.00 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Social Functioning: Change at Cycle 5 Week 24: number analyzed (Participants) | 1
  Social Functioning: Change at Cycle 5 Week 24 | 10.00 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Social Functioning: Change at Cycle 6 Week 12: number analyzed (Participants) | 1
  Social Functioning: Change at Cycle 6 Week 12 | 10.00 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Social Functioning: Change at Cycle 6 Week 24: number analyzed (Participants) | 0
  School Functioning: Change at Cycle 1 Week 12 | 5.67 (19.445)
  School Functioning: Change at Cycle 1 Week 24 | 2.00 (20.160)
  School Functioning: Change at Cycle 2 Week 12: number analyzed (Participants) | 12
  School Functioning: Change at Cycle 2 Week 12 | -5.00 (24.027)
  School Functioning: Change at Cycle 2 Week 24: number analyzed (Participants) | 12
  School Functioning: Change at Cycle 2 Week 24 | 8.75 (16.394)
  School Functioning: Change at Cycle 3 Week 12: number analyzed (Participants) | 11
  School Functioning: Change at Cycle 3 Week 12 | 3.64 (23.355)
  School Functioning: Change at Cycle 3 Week 24: number analyzed (Participants) | 9
  School Functioning: Change at Cycle 3 Week 24 | -3.33 (22.500)
  School Functioning: Change at Cycle 4 Week 12: number analyzed (Participants) | 9
  School Functioning: Change at Cycle 4 Week 12 | 0.00 (15.000)
  School Functioning: Change at Cycle 4 Week 24: number analyzed (Participants) | 7
  School Functioning: Change at Cycle 4 Week 24 | 13.57 (8.018)
  School Functioning: Change at Cycle 5 Week 12: number analyzed (Participants) | 5
  School Functioning: Change at Cycle 5 Week 12 | 15.00 (11.180)
  School Functioning: Change at Cycle 5 Week 24: number analyzed (Participants) | 4
  School Functioning: Change at Cycle 5 Week 24 | 18.75 (8.539)
  School Functioning: Change at Cycle 6 Week 12: number analyzed (Participants) | 4
  School Functioning: Change at Cycle 6 Week 12 | 13.75 (4.787)
  School Functioning: Change at Cycle 6 Week 24: number analyzed (Participants) | 1
  School Functioning: Change at Cycle 6 Week 24 | 20.00 (NA) — Standard deviation could not be calculated because single participant was analyzed.

34. Other Pre Specified Outcome: Change From Baseline In Pediatric Quality of Life Inventory (PedsQL) Generic Core Scale (GCS) Score at End of Last NTT Period During the NTT Periods in Prospective Study Period
Description: as for outcome 33
Time Frame: Baseline (from the beginning of the prospective study period), End of Last NTT period (up to Week 120)
Population: Safety population included all enrolled participants who provided informed consent for the prospective portion and met all the inclusion criteria. Data was not collected and analyzed at this time point, for this respective arms.
Arm/Group | Prospective TED/NTT Group | Prospective TED/TED Group
Number analyzed (Participants) | 0 | 0

35. Other Pre Specified Outcome: Change From Baseline In Pediatric Quality of Life Inventory (PedsQL) Family Impact Module Total Score at Week 12 and 24 of Each Treatment Cycle During the Teduglutide Treatment Periods of Prospective Study Period
Description: PedsQL Family Impact Module was composed of 36 items comprising Physical Functioning (6 items), Emotional Functioning (5 items), Social Functioning (4 items), Cognitive Functioning (5 items), Communication (3 items), Worry (5 items), Daily Activities (3 items) and Family Relationships (5 items). Total score was calculated as the sum of all the items over the number of items answered on all the scales. Scores are transformed on a scale from 0 to 100 were 0=100, 1=75, 2=50, 3=25, and 4=0. Higher scores indicate improved quality of life.
Time Frame: Baseline (from the beginning of the prospective study period), Week 12 and 24 of Cycles 1 to 6
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Prospective TED/TED Group
Number analyzed (Participants) | 19
Score on a scale
  Change at Cycle 1 Week 12: number analyzed (Participants) | 18
  Change at Cycle 1 Week 12 | 1.39 (15.742)
  Change at Cycle 1 Week 24 | 1.56 (13.372)
  Change at Cycle 2 Week 12: number analyzed (Participants) | 15
  Change at Cycle 2 Week 12 | 0.10 (13.622)
  Change at Cycle 2 Week 24: number analyzed (Participants) | 16
  Change at Cycle 2 Week 24 | 1.90 (11.664)
  Change at Cycle 3 Week 12: number analyzed (Participants) | 13
  Change at Cycle 3 Week 12 | 2.72 (15.051)
  Change at Cycle 3 Week 24: number analyzed (Participants) | 11
  Change at Cycle 3 Week 24 | 3.90 (16.018)
  Change at Cycle 4 Week 12: number analyzed (Participants) | 10
  Change at Cycle 4 Week 12 | 2.14 (20.762)
  Change at Cycle 4 Week 24: number analyzed (Participants) | 9
  Change at Cycle 4 Week 24 | 4.66 (23.546)
  Change at Cycle 5 Week 12: number analyzed (Participants) | 8
  Change at Cycle 5 Week 12 | 0.11 (14.105)
  Change at Cycle 5 Week 24: number analyzed (Participants) | 6
  Change at Cycle 5 Week 24 | 2.23 (16.099)
  Change at Cycle 6 Week 12: number analyzed (Participants) | 4
  Change at Cycle 6 Week 12 | 5.13 (18.084)
  Change at Cycle 6 Week 24: number analyzed (Participants) | 1
  Change at Cycle 6 Week 24 | -17.86 (NA) — Standard deviation could not be calculated because single participant was analyzed.

36. Other Pre Specified Outcome: Change From Baseline In Pediatric Quality of Life Inventory (PedsQL) Family Impact Module Total Score at End of Last NTT Period During the NTT Periods in Prospective Study Period
Description: as for outcome 35
Time Frame: Baseline (from the beginning of to the end the prospective study period), End of Last NTT period (up to Week 120)
Population: as for outcome 34
Arm/Group | Prospective TED/NTT Group | Prospective TED/TED Group
Number analyzed (Participants) | 0 | 0

37. Other Pre Specified Outcome: Change From Baseline In Pediatric Quality of Life Inventory (PedsQL) Gastrointestinal Symptoms Module at Week 12 and 24 of Each Treatment Cycle During the Teduglutide Treatment Periods of Prospective Study Period
Description: PedsQL GI symptoms module was composed of 58 items, comprised of 10 different symptom scales that assess gastrointestinal symptom-related quality of life: food and drink limits, trouble swallowing, heartburn and reflux, nausea and vomiting, gas and bloating, constipation, blood in poop, and diarrhea. Only the scales of food and drink limits (6 items) and diarrhea (7 items) was used in this study. Subscale score was calculated as the sum of the items over the number of items answered in the scale. Scores are transformed on a scale from 0 to 100 were 0=100, 1=75, 2=50, 3=25, and 4=0. Higher scores indicate improved quality of life.
Time Frame: Baseline (from the beginning of the prospective study period), Week 12 and 24 of Cycles 1 to 6
Population: Safety population included all enrolled participants who provided informed consent for the prospective portion and met all the inclusion criteria. Here, overall number of participants analyzed refer to the participants evaluable for this outcome measure and number analyzed refer to participants evaluable for this outcome at at specific time point at specific time point. Data for this outcome was not planned to be collected and analyzed in prospective TED/NTT group.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Prospective TED/TED Group
Number analyzed (Participants) | 19
Score on a scale
  Food and Drink Limits: Change at Cycle 1 Week 12: number analyzed (Participants) | 18
  Food and Drink Limits: Change at Cycle 1 Week 12 | -2.08 (30.460)
  Food and Drink Limits: Change at Cycle 1 Week 24 | -7.06 (27.524)
  Food and Drink Limits: Change at Cycle 2 Week 12: number analyzed (Participants) | 15
  Food and Drink Limits: Change at Cycle 2 Week 12 | -0.83 (29.723)
  Food and Drink Limits: Change at Cycle 2 Week 24: number analyzed (Participants) | 17
  Food and Drink Limits: Change at Cycle 2 Week 24 | 9.31 (26.292)
  Food and Drink Limits: Change at Cycle 3 Week 12: number analyzed (Participants) | 14
  Food and Drink Limits: Change at Cycle 3 Week 12 | 1.19 (35.784)
  Food and Drink Limits: Change at Cycle 3 Week 24: number analyzed (Participants) | 11
  Food and Drink Limits: Change at Cycle 3 Week 24 | -0.08 (29.511)
  Food and Drink Limits: Change at Cycle 4 Week 12: number analyzed (Participants) | 9
  Food and Drink Limits: Change at Cycle 4 Week 12 | -4.63 (33.750)
  Food and Drink Limits: Change at Cycle 4 Week 24: number analyzed (Participants) | 8
  Food and Drink Limits: Change at Cycle 4 Week 24 | 1.04 (35.895)
  Food and Drink Limits: Change at Cycle 5 Week 12: number analyzed (Participants) | 7
  Food and Drink Limits: Change at Cycle 5 Week 12 | 1.19 (21.343)
  Food and Drink Limits: Change at Cycle 5 Week 24: number analyzed (Participants) | 6
  Food and Drink Limits: Change at Cycle 5 Week 24 | -17.36 (44.986)
  Food and Drink Limits: Change at Cycle 6 Week 12: number analyzed (Participants) | 3
  Food and Drink Limits: Change at Cycle 6 Week 12 | -1.39 (30.142)
  Food and Drink Limits: Change at Cycle 6 Week 24: number analyzed (Participants) | 1
  Food and Drink Limits: Change at Cycle 6 Week 24 | -45.83 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Diarrhea: Change at Cycle 1 Week 12: number analyzed (Participants) | 18
  Diarrhea: Change at Cycle 1 Week 12 | 7.79 (23.137)
  Diarrhea: Change at Cycle 1 Week 24: number analyzed (Participants) | 18
  Diarrhea: Change at Cycle 1 Week 24 | 9.33 (23.279)
  Diarrhea: Change at Cycle 2 Week 12: number analyzed (Participants) | 15
  Diarrhea: Change at Cycle 2 Week 12 | 5.48 (15.144)
  Diarrhea: Change at Cycle 2 Week 24: number analyzed (Participants) | 17
  Diarrhea: Change at Cycle 2 Week 24 | 6.72 (19.880)
  Diarrhea: Change at Cycle 3 Week 12: number analyzed (Participants) | 14
  Diarrhea: Change at Cycle 3 Week 12 | 13.27 (22.124)
  Diarrhea: Change at Cycle 3 Week 24: number analyzed (Participants) | 11
  Diarrhea: Change at Cycle 3 Week 24 | 5.19 (21.569)
  Diarrhea: Change at Cycle 4 Week 12: number analyzed (Participants) | 9
  Diarrhea: Change at Cycle 4 Week 12 | 9.13 (18.653)
  Diarrhea: Change at Cycle 4 Week 24: number analyzed (Participants) | 8
  Diarrhea: Change at Cycle 4 Week 24 | 12.95 (26.448)
  Diarrhea: Change at Cycle 5 Week 12: number analyzed (Participants) | 7
  Diarrhea: Change at Cycle 5 Week 12 | 10.71 (23.237)
  Diarrhea: Change at Cycle 5 Week 24: number analyzed (Participants) | 6
  Diarrhea: Change at Cycle 5 Week 24 | 8.33 (30.612)
  Diarrhea: Change at Cycle 6 Week 12: number analyzed (Participants) | 3
  Diarrhea: Change at Cycle 6 Week 12 | 5.95 (22.961)
  Diarrhea: Change at Cycle 6 Week 24: number analyzed (Participants) | 1
  Diarrhea: Change at Cycle 6 Week 24 | -7.14 (NA) — Standard deviation could not be calculated because single participant was analyzed.

38. Other Pre Specified Outcome: Change From Baseline In Pediatric Quality of Life Inventory (PedsQL) Gastrointestinal Symptoms Module at End of Last NTT Period During the NTT Periods in Prospective Study Period
Description: as for outcome 37
Time Frame: Baseline (from the beginning of the prospective study period), End of Last NTT period (up to Week 120)
Population: as for outcome 34
Arm/Group | Prospective TED/NTT Group | Prospective TED/TED Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of screening up to end of the study (up to 168 weeks)
Arm/Group | Retrospective TED/NTT Group | Retrospective TED/TED Group | Prospective TED/NTT Group | Prospective TED/TED Group
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/5 | 0/5 | 0/19
Serious Adverse Events (participants affected / at risk) | 23/24 | 4/5 | 3/5 | 17/19
Other Adverse Events (participants affected / at risk) | 1/24 | 1/5 | 4/5 | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Retrospective TED/NTT Group (N=24) | Retrospective TED/TED Group (N=5) | Prospective TED/NTT Group (N=5) | Prospective TED/TED Group (N=19)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Congenital megacolon (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (6)
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Short-bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Complication associated with device (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperpyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 14 (31) | 3 (6) | 0 (0) | 7 (12)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 17 (33) | 2 (6) | 1 (1) | 9 (13)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Enterococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Influenza (Infections and infestations) | 5 (5) | 0 (0) | 0 (0) | 4 (4)
Metapneumovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Micrococcus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rotavirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Viral pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anastomotic ulcer (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza A virus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (4)
Feeding intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Weight gain poor (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Device breakage (Product Issues) | 6 (8) | 1 (1) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device failure (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device malfunction (Product Issues) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter management (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Central venous catheterisation (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Superior vena cava occlusion (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Retrospective TED/NTT Group (N=24) | Retrospective TED/TED Group (N=5) | Prospective TED/NTT Group (N=5) | Prospective TED/TED Group (N=19)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 3 (7)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Middle ear effusion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (4) | 7 (22)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (7)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (10)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Faecal volume increased (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastroenteritis eosinophilic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (7)
Oral mucosal erythema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Perianal erythema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post-tussive vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal discharge (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (8)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 10 (55)
Administration site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ill-defined disorder (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Medical device site irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Secretion discharge (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Croup infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Lyme disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (7)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (5) | 7 (18)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (5)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Medication error (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacterial test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Blood iron decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 5 (6)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal stoma output increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematocrit decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymph node palpable (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Occult blood positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serum ferritin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Streptococcus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin A decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
pH urine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (16)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (6)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device leakage (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (10)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nodular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2019-10-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT02949362/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-16): https://cdn.clinicaltrials.gov/large-docs/62/NCT02949362/SAP_001.pdf